CLINICAL TRIAL: NCT06142500
Title: WEST-KOaST Study: WES (Whole Exome Sequencing) Analysis of Testicular Cancer Patientsand Their First-degree Family Members
Brief Title: WEST-KOaST Study: WES Analysis of Testicular Cancer Patientsand Their First-degree Family Members
Acronym: West-KOaSt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: West KOaSt
Record Dates: First submitted 2023-10-09; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Testicular Cancer
Keywords: testicular cancer; cancer; familiarity; genetic; male infertility
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms; Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with testicular cancer (Experimental): Patient with testicular cancer
  Interventions: Genetic: Analysis of biological samples of saliva from testicular cancer patients and from their first-degree family members
- First-degree family members of patients with testicular cancer (Active Comparator): First-degree family members of patients with testicular cancer
  Interventions: Genetic: Analysis of biological samples of saliva from testicular cancer patients and from their first-degree family members

INTERVENTIONS:
Genetic: Analysis of biological samples of saliva from testicular cancer patients and from their first-degree family members — The project aims to collect biological samples of saliva from testicular cancer patients and from their first-degree family members; demographic-clinical variables will be also collected in order to draft a comprehensive panel of genes and gene modifications related to the testicular cancer, combining this survey with a very detailed descprition of this cohort of patient in terms of clinical features and quality of life

SUMMARY:
The project aims to identify the possible risk factors regarding the onset of the disease and to evaluate genes and gene modifications responsible for the onset od testicular cancer.

DETAILED DESCRIPTION:
Testicular tumor represents a relatively rare disease that hit young-adults men. It represents 1% of all male cancers and 5% of all urological male tumors. Its incidence grow year by year. In the field of the oncological research, the lack of knowledge about genes related to this disease represent a very relevant clinical question. For this reason this project aims to collect biological samples of saliva from testicular cancer patients and from their first-degree family members; demographic-clinical variables will be also collected in order to draft a comprehensive panel of genes and gene modifications related to the testicular cancer, combining this survey with a very detailed description of this cohort of patient in terms of clinical features and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male testicular cancer patients with an age > 18 and < 90
* First degree family members of Male testicular cancer patients with an age > 18 and < 90
* Ability to read and sign the informed consent
* Diagnosis of testicular cancer for the experimental group

Exclusion Criteria:

* Female for the experimental group
* Second degree family members of Male testicular cancer patients
* People with an age < 18 and > 90
* Diagnosis different from testicular cancer for the experimental group Incapacity to read and sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Saliva biological sample | Baseline
  Saliva biological samples will be collected from both patients with testicular cancer and their first-degree family members trough a buccal swab, that will be analysed with a whole exome sequencing (WES) in order to explore panel of genes

SECONDARY OUTCOMES:
Demographic-clinical variables | Baseline
  Demographic and clinical variables will be collected from the interview with the physician: 1)Age of the subject; 2. Age at diagnosis; 3. Ethnicity; 4.BMI; 5. Lifestyle (smoking, diet, alcohol, physical activity…); 6. Histotype of the neoplasm; 7; Nodule Size; Presence of embryonal carcinoma > 50%; 8. Percentage of necrosis present; 9. Basic pharmacological therapy; 10. Chemo/radiotherapy;

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele

IPD SHARING:
Plan to Share IPD: No